CLINICAL TRIAL: NCT00807677
Title: A Phase 1 Dose Escalation Study of TAK-901 in Subjects With Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-901_101
Record Dates: First submitted 2008-12-10; First posted 2008-12-12 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Chronic Lymphocytic Leukemia; Multiple Myeloma; Waldenstrom's Macroglobulinemia; Myelodysplastic Syndrome; Philadelphia Chromosome-negative CML; Myeloid Metaplasia; Myelofibrosis; Advanced Polycythemia; Non-Hodgkins Lymphoma
Keywords: Chronic myelogenous leukemia (CML) in chronic phase, accelerated phase, or blast crisis; Intermediate or high risk myelodysplastic syndrome; Philadelphia chromosome-negative CML (including blast phase); All subtypes of myeloid metaplasia with myelofibrosis; advanced polycythemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia; Myelodysplastic Syndromes; Primary Myelofibrosis; Lymphoma, Non-Hodgkin; Blast Crisis | interventions — TAK-901

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): TAK-901
  Interventions: Drug: TAK-901

INTERVENTIONS:
Drug: TAK-901 — TAK-901 will be administered via IV infusion over a 3-hour period on Days 1,4,8,11,15,18,22, and 25 of each 28-day cycle.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of TAK-901 in subjects with advanced hematological malignancies, and to further assess the safety and tolerability of TAK-901 at or below the MTD in an expanded cohort of subjects in order to select a dose for future studies.

ELIGIBILITY:
Main Inclusion Criteria:

1. The subject has one of the following confirmed diseases that is refractory to or relapsed from established therapies. Note: A subject with one of these disease who is intolerant (as defined in the protocol) to established therapies is also allowed:

   1. Acute myelogenous leukemia
   2. Acute lymphoblastic leukemia
   3. Chronic myelogenous leukemia (CML) (chronic phase, accelerated phase, or blast crisis)
   4. Chronic lymphocytic leukemia
   5. Multiple myeloma
   6. Waldenstrom's macroglobulinemia
   7. Intermediate or high risk myelodysplastic syndrome
   8. One of the following myeloproliferative disorders:

      * Philadelphia chromosome-negative CML (including blast phase).
      * All subtypes of myeloid metaplasia with myelofibrosis.
      * Advanced polycythemia vera in the spent phase (ie, presence of anemia).
   9. Non-Hodgkins lymphoma
2. The interval between the last prior treatment and the start of study drug administration is at least 30 days for radiotherapy, at least 14 days for cytotoxic chemotherapy (42 days for nitrosureas or mitomycin C), and at least 5 half-lives for noncytotoxic agents. The only exception is hydroxyurea, which can be used prior to starting study drug and during Cycle 1, as defined in the protocol.
3. For subjects with prior autologous bone marrow or peripheral blood stem cell transplantation, the interval between transplant and the start of study drug administration is at least 30 days.
4. For subjects with prior allogeneic bone marrow or peripheral blood stem cell transplantation, the interval between transplant and the start of study drug administration is at least 90 days.
5. If taking steroids chronically, the subject has been receiving a stable steroid dose for at least 21 days prior to the start of study drug administration, and the daily steroid dose does not exceed the equivalent of 20 mg prednisone.
6. The subject is aged 18 years or older.
7. The subject weighs at least 45 kg.
8. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
9. The subject has adequate liver and kidney function.
10. The subject has adequate heart function (left ventricular ejection fraction ≥ 50%).

Main Exclusion Criteria:

Any subject who meets any of the following criteria will not qualify for entry into the study:

1. The subject has a platelet count (untransfused) < 50,000/mm3 and/or an absolute neutrophil count < 1000/mm3 that is not caused by the underlying disease infiltrating the bone marrow.
2. The subject has evidence of active malignancy in the central nervous system (CNS)or has had CNS involvement documented within the past 90 days. Subjects who are receiving maintenance intrathecal chemotherapy for previous CNS involvement but have no current evidence of disease are allowed if the CNS involvement was documented more than 90 days ago.
3. The subject has any evidence of acute or chronic graft versus host disease.
4. The subject has a history of hypersensitivity or allergic reactions attributed to compounds of similar chemical composition to TAK-901 or its excipient, Captisol.
5. The subject is pregnant or lactating.
6. The subject has had a myocardial infarction, cerebrovascular accident, transient ischemic attack, clinically significant ventricular arrhythmia, or pulmonary embolus within 6 months prior to the start of study drug administration.
7. The subject's electrocardiogram demonstrates an abnormal QT interval , as defined by the protocol.
8. The subject requires dialysis.
9. The subject is on systemic anticoagulation therapy.
10. The subject has an uncontrolled intercurrent illness as defined in the protocol.
11. The subject is known to have human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
12. The subject has a currently active second malignancy other than nonmelanoma skin cancer or in situ carcinoma of the cervix. A malignancy is considered to be currently active if the subject is receiving ongoing therapy or has been in remission for less than 2 years prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose(MTD)of TAK-901 in subjects with advanced hematologic malignancies. | Duration of the study
To further assess the safety and tolerability of TAK-901 at or below the MTD in an expanded cohort of subjects in order to select a dose for future studies. | Duration of study

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic profile of TAK-901 and its primary metabolite (M-I). | Duration of the study
To make a preliminary assessment of the clinical activity of TAK-901. | Duration of therapy
To make a preliminary assessment of the effects of TAK-901 on pharmacodynamic biomarkers. | Duration of therapy
To make a preliminary assessment of the association between selected genetic markers and TAK-901 response and/or pharmacokinetic parameters. | Duration of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States